CLINICAL TRIAL: NCT06981325
Title: Evaluation of Efficacy and Safety of Cemiplimab as First Line Treatment for Advanced Basal Cell Carcinoma (CEMI-first) - An Open Label, Single Arm, Prospective Phase II Trial of the DeCOG Network
Brief Title: Evaluation of Efficacy and Safety of Cemiplimab as First Line Treatment for Advanced Basal Cell Carcinoma (BCC) Patients
Acronym: CEMI-first
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Skin Cancer Center Minden, Department of Dermatology, Johannes-Wesling-Klinikum Minden (Unknown); Translational Skin Cancer Research, University Duisburg-Essen (Unknown); Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEMI-first
Record Dates: First submitted 2025-03-06; First posted 2025-05-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Basal Cell Carcinoma (BCC); First Line Treatment
Keywords: BCC; Skin Cancer; Basal Cell Carcinoma; anti-PD-1 monoclonal antibody; HHI naïve; Cemiplimab
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Intervention Model Description: Clinical trial with a single arm, all eligible patients will receive Cemiplimab 350 mg (i.v.) on day 1 of every 21 cycle for up to 12 months (max. 17 cycles) or until intolerable toxicity or disease progression, whatever occurs first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cemiplimab - Single Arm (Experimental): Single Arm with Cemiplimab 350 mg i.v. on day 1 of every 21 days cycle for up to 12 months (max. 17 cycles).
  Interventions: Drug: Cemiplimab

INTERVENTIONS:
Drug: Cemiplimab — Cemiplimab 350 mg i.v. on day 1 of every 21 days cycle for up to 12 months (max. 17 cycles).
  Other Names: LIBTAYO

SUMMARY:
The study is an open-label, singel arm, prospective, multicenter phase II trial evaluating the efficacy and safety of Cemiplimab when applied as first-line therapy in patients with locally advanced basal cell carcinoma (BCC), which were not pretreated with hedgehog inhibitors (HHI).

DETAILED DESCRIPTION:
The present study is an explorative, investigator-initatied, single-arm, multicentre phase II trial. Patients with locally advanced BCC without pretreatment with hedgehog inhibitors such as vismodegib and sonidegib will receive Cemiplimab (350 mg, i.v.) at day 1 of each 21 days cycle for up to 12 months (max. 17 cycles) or until intolerable toxicity or disease progression, whatever occurs first. All patients will be followed up until death or for up to 12 months after last patient last application of Cemiplimab. The treatment response will be assessed every 12 weeks (± 7 days) during the treatment and the follow up phase. In addition, tumor samples will be collected and used for translational research providing the basis for the establishment of potential biomarkers correlating with the efficacy of Cemiplimab. The primary objective of this study is to evaluate the efficacy of Cemiplimab when applied as first-line treatment in advanced, HHI naïve BCC measured by objective response rate (ORR) after 6 months of treatment. Secondary objective is to evaluate the safety and tolerability of Cemiplimab as first-line treatment in advanced BCC.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form available
2. Patient* 18 years or older at time of signing informed consent form
3. Centrally confirmed histological diagnosis of BCC

   NOTE: Tumor tissue to be sent to Central Pathology during screening procedure:
   * Formalin-fixed, parrafin-embedded (FFPE) tumor specimen in a paraffin block (preferred) OR
   * approximately 10 sections (5µm thickness) on uncoated slides and 10 sections (3µm thickness) on Superfrost Ultra slides containing unstained, freshly cut, serial sections to be submitted along with associated pathology report (please refer to section 11.1.1 for details)
4. Locally advanced stage without distant metastases, not amenable for surgery or radiotherapy or surgery/radiotherapy contraindicated or refused by patient (as evidenced in source data)
5. Expected survival of at least 6 months
6. ECOG performance status 0 or 1
7. Adequate laboratory parameters particularly for the blood count, renal and liver function parameters.

   1. Absolute number of neutrophils ≥ 1.5 x 109/L
   2. Platelets ≥ 75 x 109/L
   3. Hemoglobin ≥ 9 g/dL
   4. Total bilirubin ≤ 1.5 times the upper limit of normal (ULN), (patients with Gilbert´s Disease and total bilirubin up to 3x ULN may be eligible after approval from trial's medical expert)
   5. AST (SGOT) and ALT (SGPT) ≤ 3x ULN
   6. AP ≤ 2.5x ULN
   7. Serum creatinine ≤ 2x ULN or creatinine clearance ≥ 40 mL/min
8. Absence of other severe comorbidities
9. Resolution of any acute, clinically significant treatment-related adverse events from prior therapy/procedure to Grade ≤ 1 prior to study entry, with the exception of alopecia.
10. Negative serum pregnancy test done less than or equal to 7 days prior to enrollment, for females of childbearing potential only.
11. Sexually active women of childbearing potential (WOCBP) and men with WOCBP partners must be prepared to use suitable contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 6 months after the last dose of Cemiplimab

    * There are no data that indicate special gender distribution. Therefore, patients will be enrolled in the study gender-independently

Exclusion Criteria:

1. Pretreatment with systemic immunotherapy (such as PD-1/PD-L1 or CTL4) or targeted therapy (such as hedgehog inhibitor) NOTE: Prior treatment with imiquimod or other topical or intralesional immune modulators will not be exclusionary
2. Any other non-radiation anti-cancer therapy (e.g. imiquimod, photodynamic therapy; neither investigational nor standard of care) within 30 days (from date of last administration) of initial Cemiplimab administration or if planned during the study duration
3. Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required systemic immunosuppressive therapy, excluding: vitiligo, childhood asthma that has resolved, type 1 diabetes, residual hypothyroidism requiring only hormone replacement, or psoriasis that does not require systemic treatment
4. Other neoplasia, in particular hematologic diseases that might impair immune response, such as chronic lymphocytic leukemia, myelodysplastic or myeloproliferative disease and patients with Gorlin-Goltz syndrom
5. Immunosuppressive corticosteroid doses (> 10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of Cemiplimab NOTE: Patients who require brief courses of steroids (e.g., as prophylaxis for imaging studies due to hypersensitivity to contrast agents) are eligible for participation. Furthermore, patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or replacement in case of adrenal or hypophysis insufficiency are eligible for participation.
6. Known allergic/hypersensitive reaction to the study drug and any of its excipients or history of documented allergic/hypersensitive reactions to antibody treatments
7. Active infection requiring systemic therapy, including uncontrolled HIV, HBV and HCV infection or diagnosis of immunodeficiency.

   NOTE: Patients are eligible if:
   * Patients have controlled HIV infection with CD4 counts is > 350 cells/µL and viral load is undectable [HIV RNA PCR]
   * Patients positive for HBV surface antigen have controlled HBV infection receiving anti-viral therapy and with undectable serum viral load [HBV DNA PCR]. Patients must remain on anti-viral therapy for at least 6 months after last dose of Cemiplimab
   * Patients positive for HCV antibody have controlled HCV infection with undectable viral load [HCV RNA PCR]
8. History of pneumonitis within the last 3 years
9. Patients with history of solid organ transplant (patients with prior corneal transplants may be allowed to enroll after discussion with and approval from the Lead Investigator)
10. Comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
11. Receipt of live vaccines (including attenuated) within 30 days of first administration of Cemiplimab
12. Pregnancy or lactation period.
13. Medical or psychological conditions that would not permit the patient to complete the study or sign informed consent.
14. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
15. Legal incapacity or limited legal capacity.
16. On-treatment participation in another clinical trial in the period 30 days prior to start of the study treatment and during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) at six months | 24 months
  ORR@6months, defined as the rate of patients assessed with complete or partial response (CR or PR) according to ERIVANCE-like criteria as best overall response, relative to the total number of patients as evaluated 6 months after treatment allocation.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 42 months
  rate of patients assessed with complete or partial response (CR or PR) as best overall response, relative to the total number of patients.
Progression Free Survival (PFS) | 42 months
  time from date of allocation to treatment to the date of the first objectively documented tumor progression, as determined by investigators, or death due to any cause.
Duration of Response (DoR) | 42 months
  length of time from initial response (CR/PR) to first objectively documented progression or death.
Overall Survival (OS) | 42 months
  time from date of allocation to treatment until the date of death from any cause
Time to next systemic treatment (TTNsT) | 42 months
  time from date of allocation to treatment to initiation of the next line of systemic therapy
Safety (AEs and SAEs) | 42 months
  Incidence of adverse events and serious adverse events
AE severity | 42 months
  Severity of adverse events by CTCAE v5.0 grade
Safety (AEs) | 42 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

OTHER OUTCOMES:
Determination of molecular biomarkers and their correlation with objective response rate (ORR) | 42 months
  Biosamples will be used for determination of molecular biomarkers and their correlation with objective response rate (ORR) by assessing e.g., gene expression signatures, tumor mutational burden including mutational signatures as well as morphological and cellular characteristics of the tumor microenvironment.

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr. med., Study Director — Institut für Klinische Krebsforschung IKF GmbH; Ralf Gutzmer, Prof. Dr. med., Principal Investigator — Johannes Wesling Klinikum Minden
Locations (7):
- Germany (7):
  - Helios Klinikum Erfurt, Erfurt
  - Universitätsklinikum Erlangen, Erlangen
  - Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
  - Universitätsklinikum Leipzig, Leipzig
  - Johannes Wesling Klinikum, Minden
  - Helios Klinikum Oberhausen, Oberhausen
  - Universitätsklinikum Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.